CLINICAL TRIAL: NCT01147939
Title: A Randomised Phase III Study of Elacytarabine vs. Investigator's Choice in Patients With Late Stage Acute Myeloid Leukaemia
Brief Title: Study of Elacytarabine Versus Investigator's Choice in Patients With Late Stage Acute Myeloid Leukaemia (AML)
Acronym: CLAVELA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP4055-306
Record Dates: First submitted 2010-04-14; First posted 2010-06-22 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukaemia; AML; Haematology; Investigator's Choice; Elacytarabine; Refractory or relapsed AML; Phase III; Randomized; CLAVELA; CP4055-306; Elacyt
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 5'-oleoyl cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elacytarabine (Experimental)
  Interventions: Drug: Elacytarabine
- Investigator's Choice (Active Comparator)
  Interventions: Drug: Investigator's Choice

INTERVENTIONS:
Drug: Elacytarabine — Elacytarabine 2000 mg/m2/d administered as a continuous intravenous infusion (CIV) in a d 1-5 q3w cycle.
  Arms: Elacytarabine
Drug: Investigator's Choice — E.g. cytarabine single agent/combinations, hypomethylating agents, best supportive care (BSC)
  Arms: Investigator's Choice

SUMMARY:
The purpose of the study is to assess the efficacy and safety of elacytarabine versus investigator's choice treatment in patients with relapsed or refractory acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
The study investigates the new nucleoside analogue derivative, elacytarabine, as treatment for patients with relapsed or refractory Acute Myeloid Leukemia (AML). To be included in the study, patients must have failed to respond to two or three different therapies for AML, or have obtained remission but then relapsed within a relatively short period of time. Patients of age ≥ 65 with adverse cytogenetics can be included in the study after having received one and up to three previous induction/re-induction therapies.

Elacytarabine is an investigational drug which is not commercially available. It is the elaidic acid ester derivative of cytarabine. Cytarabine is routinely used in the treatment of patients with AML. A substantial portion of AML patients have a deficient uptake of cytarabine, often explained by lack of a transport protein (hENT1) in the leukemic cell membrane. Due to the elaidic acid (a naturally occurring fatty acid), cellular uptake of elacytarabine is independent of this transport protein.

Patients included in the study will be randomized to elacytarabine or control treatment. Since there is no standard therapy for relapsed or refractory AML, there is a list of 7 control treatments and the investigator has to choose one that is locked before randomization.

Elacytarabine is given as a continuous infusion over five days, followed by a rest period of minimum two weeks. Investigator's choice treatment is given according to the specific routine.

After each course response evaluation and a decision on further treatment will be made.

Repeated courses of elacytarabine and control treatment might be needed to attain and/or maintain complete remission or clinical benefit.

After the end of study treatment, all patients will be followed for relapse and survival.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Confirmed diagnosis of AML according to WHO classification (excluding acute promyelocytic leukaemia) who have received two or three previous induction/re-induction regimens or patients of age ≥ 65 with adverse cytogenetics who have received 1-3 previous induction/re-induction regimens. One of the (re-)induction regimens could be stem cell transplantation (SCT) for achievement of remission. Maintenance and consolidation (including SCT) may have been given, but are not counted as previous regimens.
* Bone marrow aspirates and/or biopsies must contain > 5 % leukaemic blast cells or patient must have biopsy-proven extramedullary AML, or patient's peripheral blood shows occurrence of leukaemic blast cells
* Patients must

  * have never attained CR or CRi (primary refractory), or
  * have failed initial induction therapy, and have attained CR or CRi after salvage therapy(ies), and then relapsed within < 6 months, or
  * have attained CR or CRi after initial induction therapy and relapsed within <12 months, and failed to respond to salvage therapy(ies), or
  * have relapsed after the latest CR or CRi within < 6 months
* Patients younger than 65 years should have received previous treatment with cytarabine
* Patients must have recovered from previous bone marrow and/or stem cell transplantation to a stage that the patient can tolerate the study treatment. There is no restriction on number of regimens or type of treatment administered for maintenance or consolidation during previous stages of the disease
* ECOG performance status (PS) of 0 - 2
* Women of child-bearing potential must have a negative serum or urine pregnancy test within 2 weeks prior to treatment start
* Male and female patients must use acceptable contraceptive methods for the duration of time on study, and males also for 3 months after the last elacytarabine dose
* Capable of understanding and complying with protocol requirements, and must be able and willing to sign a written informed consent form

Exclusion Criteria:

* A history of allergic reactions to egg. A history of allergic reactions of CTCAE grade 3 or 4 to cytarabine
* Persistent clinically significant toxicities from previous chemotherapy
* A cancer history that, according to the investigator, might confound the assessment of the study endpoints
* Known positive status for human immunodeficiency virus (HIV)
* Pregnant and nursing patients
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Impairment of hepatic or renal function to such an extent that the patient, in the opinion of the investigator, will be exposed to an excessive risk if entered into this clinical study
* Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure. Any New York Heart Association (NYHA) functional classification grade 3 or 4
* Applicable only for patients for whom an anthracycline is part of the selected control treatment: Left ventricular ejection fraction (LVEF) must be ≥ 45 % as measured by MUGA scan or 2D ECHO within 14 days prior to start of therapy. Either method is acceptable for measuring LVEF
* Applicable only for patients for whom an anthracycline is part of the selected control treatment: The patient should tolerate minimum one course of combination therapy
* Any anti-leukaemic agents within the last 3 weeks. Hydroxyurea,however, is allowed for up to 12 hours prior to study treatment
* Any investigational treatment within the last 14 days
* Any medical condition which in the opinion of the investigator places the patient at an unacceptably high risk for toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2010-06; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | Until 300 events occur
  Time from date of randomisation until the date of death

SECONDARY OUTCOMES:
Remission rate | Until 300 events occur
  * Remission rate measured by overall response rate (ORR) (i.e. complete remission (CR) and complete remission with incomplete bone marrow recovery (CRi))
  * Remission rate measured by CR
  * Remission duration analysed using cumulative incidence of relapse (CIR) measured from date of CR or CRi
Compare number of patients with adverse events (AEs) per study arm as a measure of safety and tolerability | From first dose of study treatment, until 30 days after the last dose (for each patient)
  Summaries will include rates of occurrence of any AEs, rates of AEs by system organ classification (SOC),rates of discontinuation of study treatment due to AEs.
Characterize exposure-response relationships for measures of effectiveness and toxicity | During the first course of elacytarabine

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke University Medical Center, Durham, NC, USA; Francis J Giles, MD, PhD, Study Chair — Cancer Therapy & Reseach Center at the University of Texas Health Science Center San Antonio, TX, USA
Locations (73):
- United States (23):
  - Scripps Cancer Center Clinical Research, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - UCLA School of Medicine, Division of Hematology/Oncology, Los Angeles, California
  - Rocky Mountain Blood and Bone Marrow Transplant Program, Denver, Colorado
  - Shands at the University of Florida, Gainesville, Florida
  - Winship Cancer Institute at Emory, Atlanta, Georgia
  - The Blood and Marrow Transplant Group of GA, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St. Francis Hospital and Health Center, Indianapolis, Indiana
  - University of Iowa Hopsitals, Iowa City, Iowa
  - LSU Health Sciences Center,, Shreveport, Louisiana
  - Northern New Jersey Cancer Associates, Hackensack, New Jersey
  - New York Presbyterian Hospital, Weill-Cornell Medical College, New York, New York
  - Memorial Sloan-Kettering, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Health Sciences Section on Hematology and Oncology, Winston-Salem, North Carolina
  - The Jewish Hospital, Cincinnati, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - St. Francis Hospital, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Froedtert Hospital, Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Royal North Shore Hopsital, Sydney, New South Wales
  - Alfred Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Belgium (6):
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - University Hospital Antwerp, Edegem
  - CHU Liège, Liège
  - UCL Mont-Godinne, Yvoir
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (7):
  - CHU Limoges - Hôpital Dupuytren, Limoges
  - Hopital Edouard Herriot, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint Antoine, Paris
  - CHU de Bordeaux - Hopital Haut-Leveque, Pessac
  - CHU de Toulouse - Hôpital Purpan, Toulouse
- Germany (8):
  - Charité-Campus B. Franklin Med. Klinik Haematology, Berlin
  - Evangelische Kliniken Johanniter- und Waldkrankenhaus Bonn GmbH, Bonn
  - Heinrich-Heine Universität Düsseldorf, Klinik für Hämatologie/Onkolog. und Klin. Immunologie, Düsseldorf
  - III. Medizinische Klinik und Poliklinik;Hämatologie, Onkologie und Pneumologie, Mainz
  - Universitätsklinikum Münster, Medisinische Klinik & Poliklinik A, Münster
  - Universitätsklinikum Rostock, Rostock
  - Robert-Bosch-Krankenhaus, Abt.Hämatologie,Onkologie u.Palliativmedizin, Stuttgart
  - Universitätsklinikum Ulm, Klinik für Innere Medizin III, Comprehensive Cancer Center Ulm (CCCU), Ulm
- Ireland (2):
  - St James's Hospital Dublin, Dublin
  - University Hospital Galway, Galway
- Italy (6):
  - A.O.U Careggi, Florence
  - A.O San Martino, Genova
  - Fondazione San Raffaele del Monte Tabor, Milan
  - A.O. Cardarelli, Napoli
  - Hospital S. Maria delle Croci, Ravenna
  - Fondazion Policlin T Vergata, Roma
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Oslo University Hospital, Oslo
  - St Olavs Hospital, Trondheim
- Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw, Poland
- Romania (3):
  - Fundeni Clinical Institute "Stefan Berceanu" Center for Hematology and Bone Marrow Transplant, Bucharest
  - Oncology Institute ,,Ion Chiricuta" Cluj Napoca , Hematology dept., Cluj-Napoca
  - St. Spiridon" University Hospital, Hematology Department, Iași
- Spain (6):
  - Hospital de Navarra, Pamplona, Spain
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitari Son Dureta, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario La Fé, Servicio de Hematología, Valencia
- United Kingdom (3):
  - Gartnavel General Hospital: Beatson WOS Cancer Centre, Glasgow, Scotland
  - Bristol Haematology and Oncology Centre, Bristol
  - Christie Hospital, Haematology and Transplant Day Unit, Manchester

REFERENCES:
- [Derived] Roboz GJ, Rosenblat T, Arellano M, Gobbi M, Altman JK, Montesinos P, O'Connell C, Solomon SR, Pigneux A, Vey N, Hills R, Jacobsen TF, Gianella-Borradori A, Foss O, Vetrhusand S, Giles FJ. International randomized phase III study of elacytarabine versus investigator choice in patients with relapsed/refractory acute myeloid leukemia. J Clin Oncol. 2014 Jun 20;32(18):1919-26. doi: 10.1200/JCO.2013.52.8562. Epub 2014 May 19. PMID 24841975
- See also: Related Info — http://www.clavispharma.com